CLINICAL TRIAL: NCT01490489
Title: EG-VEGF (Endocrine Gland-derived Vascular Endothelial Growth Factor) in Normal and Pathological Pregnancies: Potential Marker of Pre-eclampsia and / or Intrauterine Growth Restriction
Brief Title: EG-VEGF : Potential Marker of Pre-eclampsia and / or Intrauterine Growth Restriction
Acronym: EGEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C09-43; 2009-A01304-53 (Registry Identifier: IDRCB)
Record Dates: First submitted 2011-12-08; First posted 2011-12-13 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2021-08

CONDITIONS: Pre-eclampsia; Intra-uterine Growth Retardation
Keywords: EG-VEGF; Endocrine Gland-derived Vascular Endothelial Growth Factor; Pre-eclampsia; intra-uterine growth retardation; prognosis
MeSH Terms: conditions — Pre-Eclampsia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregnent women with blood sample (Other)
  Interventions: Other: blood sample and doppler Ultrasound of uterine arteries

INTERVENTIONS:
Other: blood sample and doppler Ultrasound of uterine arteries — * 36 ml of blood samples (serum and plasma) will be collected
  * After a bed rest supine for 15 minutes, ultrasound Doppler from each of the uterine arteries will be performed to search for Notch

SUMMARY:
The purpose of this study is to assess the potential prognostic value of seric concentrations of EG-VEGF for Pre-eclampsia and/or intrauterine growth restriction and will allow checking whether plasma levels of EG-VEGF at 14-18 weeks of gestation could be proposed as prognostic marker for preeclampsia.

DETAILED DESCRIPTION:
Successful human placentation depends on adequate transformation of the uteroplacental vasculature by extravillous trophoblast (EVT) following proliferation, migration, and invasion of these cells into the maternal decidua. This process of vascular remodelling rises to a peak by the end of the first trimester and declines rapidly thereafter. Poor invasion can lead to the development of pathological condition such as Pre-eclampsia (PE) and intrauterine growth restriction (IUGR). PE affects 5-6 % of pregnancies in France and causes the death of ten or so women per year. Our research project is dedicated to the comprehension of the mechanisms underlying the development of PE and to the search of gold prognostic marker of this pathology. We were particularly interested in the study of the new angiogenic factor, EG-VEGF, recently reported as new factor specific to endocrine glands including the placenta. In recent results obtained by our team, we have shown that i) placental EG-VEGF showed a peak of expression just before the establishment of the foeto-maternal circulation ii) EG-VEGF receptors, PKR1 and PKR2 were also expressed during the first trimester of pregnancy and iii) EG-VEGF expression and that of its receptor PKR1 were up-regulated by hypoxia. In our last publication "under press in JCMM" we have shown that EG-VEGF inhibits EVT migration and invasion. More importantly, we have succeeded to measure EG-VEGF circulating levels in non pregnant and in pregnant women at the three trimesters of pregnancy and showed that its highest levels (5 times the non pregnant levels) were found during the first trimester of pregnancy with a significant decrease thereafter. Furthermore, on a cohort of 19 PE patient and 21 age matched controls, we have observed a significant increase in EG-VEGF levels in the PE group. Therefore we hypothesize that EG-VEGF could play an important role in human placentation and that a persistence in its expression over the first trimester of pregnancy may contribute to the development of PE.

Based on the Doppler analysis method for the assessment of uterine artery transformation by the end of 1st trimester, we propose to search for a correlation between the circulating levels of the new angiogenic factor EG-VEGF in the sera of pregnant woman between 14 to 18 WG, and the development of PE and/or IUGR. Doppler ultrasonography is a predictive method of the pregnancy outcome at the time of the development of the disease (1st to 2nd trimester), before threatening symptoms launch (end of the 2nd to the 3rd trimester). In normal pregnancy, impedance to flow in the uterine arteries decreases with gestation as result of trophoblastic invasion of the spiral arteries and their conversion into low-resistance vessels by the end of first trimester of pregnancy. Therefore, the present study will also allow the search for a negative correlation between the level of uterine artery transformation and the level of EG-VEGF. The study will be conducted in collaboration with the Clinical centre of the Grenoble CHU Hospital (Dr JL. Cracowski). In this study we plan to include 500 pregnant pregnant women. Patients will be recruited at the time of their first ultrasonography between 11 and 13 WG and included in the study between 14 and 18 WG. For each patient a blood sample will be taken for the measurement of circulating EG-VEGF and Doppler analysis for uterine artery transformation will be performed. These results will provide information concerning the potential prognostic value of seric concentrations of EG-VEGF for PE and/or IUGR and will allow checking whether plasma levels of EG-VEGF at 14-18 weeks of gestation could be proposed as prognostic marker for preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 17 years old
* All pregnant patients enrolled before 14 SG and with singleton, irrespectively of their parity
* Pregnant woman living in the Grenoble area
* Women accepting, the participation to the study.

Exclusion Criteria:

* Inability to understand the project
* Persons deprived of their liberty by judicial or administrative decisions
* Person under legal protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2011-07-11 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-03-13 (Actual)

PRIMARY OUTCOMES:
Measure of the circulating levels of EG-VEGF in the sera of pregnant woman between 14 and 18 WG | Between 14 and 18 weeks of gestation
  Measure the circulating levels of the new angiogenic factor EG-VEGF in the sera of pregnant woman between 14 and 18 WG to determine whether EG-VEGF could represent a prognostic marker for the development of PE and/or IUGR

SECONDARY OUTCOMES:
Correlation between the level of uterine artery transformation and the level of EG-VEGF. | Between 14 and 18 week of gestation
  Correlation between the level of EG-VEGF and the level of uterine artery transformation evaluated by Doppler ultrasound.
Measure the circulating levels of other pro and/or anti-angiogenic factors | Between 14 and 18 week of gestation
  Measure the circulating levels of other pro and/or anti-angiogenic factors that could represent alternative biomarkers in the development of placental pathologies of vascular origin. As candidates, we will measure the soluble receptor of VEGF (s-flt) and Bone morphogenetic protein-9 (BMP9)
Measure the circulating levels of the new angiogenic factor EG-VEGF | Between 14 and 18 weeks of gestation
  Measure the circulating levels of the new angiogenic factor EG-VEGF in the sera of pregnant woman between 14 and 18 WG to determine whether EG-VEGF could represent a prognostic marker for the development of PE.
Measure the circulating levels of the new angiogenic factor EG-VEGF in the sera | Between 14 and 18 weeks of gestation
  Measure the circulating levels of the new angiogenic factor EG-VEGF in the sera of pregnant woman between 14 and 18 WG to determine whether EG-VEGF could represent a prognostic marker for the development of IUGR

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Hoffmann, MD/PHD, Principal Investigator — University Hospital, Grenoble; Nadia ALFAIDI, PHD, Study Director — inserm U878
Locations (1):
- Clinical investigation center of the Grenoble University Hospital, Grenoble, Isere, France